CLINICAL TRIAL: NCT07335783
Title: Results of Lunocapitate Fusion in Mangement of Scaphoid Non Union Advanced Collapse (SNAC Wrist)
Brief Title: Lunocapitate Fusion in Snac Wrist
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hany Ahmed Ali, Resident, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Snac wrist lunocapitate fusion
Record Dates: First submitted 2025-12-31; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Snac Wrist

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lunocapitate fusion (Experimental)
  Interventions: Procedure: Results of lunocapitate fusion in mangement of scaphoid non union Advanced collapse (SNAC wrist); Procedure: Lunocapitate fusion in snac wrist

INTERVENTIONS:
Procedure: Results of lunocapitate fusion in mangement of scaphoid non union Advanced collapse (SNAC wrist) — Lunocapitate fusion in snac wrist
Procedure: Lunocapitate fusion in snac wrist — Lunocapitate (LC) fusion has emerged as a promising salvage technique. By reducing the number of fusion sites compared to other procedures, it aims to achieve a higher union rate, reduce operative time, and better preserve wrist motion. However,comprehensive prospective data on its outcomes are still needed. This study will prospectively evaluate the efficacy and safety of lunocapitate fusion as a primary surgical treatment for SNAC wrist.

SUMMARY:
Scaphoid fractures are common, accounting for approximately 60-70% of all carpal bone fractures. StatPearls. Scaphoid Wrist Fracture. (2024). (A significant challenge is the high rate of missed or delayed diagnosis, which occurs in up to 30% of cases initially, often due to subtle radiographic findings). [Orthobullets - Acute Scaphoid Fractures] This is critical because 10-20% of acute scaphoid fractures are prone to nonunion even with appropriate treatment,[ResearhGate - Scaphoid Non-Union]. a risk that rises dramatically to over 80-90% if the fracture is completely untreated or missed.ResearchGate Nonunion can lead to scaphoid nonunion advanced collapse (SNAC) is a progressive and debilitating wrist disorder that arises from an untreated scaphoid fracture, leading to characteristic patterns of osteoarthritis. Surgical intervention is often required to alleviate pain and improve function.National Library Of Medicine Treatment strategies vary based on fracture timing and union status. For acute, nondisplaced fractures, non-surgical management with cast immobilization for 8-12 weeks is the standard initial approach, For displaced acute fractures or cases of established nonunion, surgical intervention is mandatory. Options include open reduction and internal fixation (ORIF) with a compression screw, often with bone grafting. In advanced stages where arthritis has developed (SNAC wrist), salvage procedures like proximal row carpectomy or limited carpal fusions are required. [Orthobullets - Scaphoid Fracture Among the available salvage procedures, lunocapitate (LC) fusion with scaphoid excision presents a compelling surgical option. This technique aims to reduce pain by eliminating the arthritic joint surfaces and stabilizing the midcarpal joint. The theoretical advantages of LC fusion include a simplified biomechanicalconstruct with fewer fusion surfaces, which may potentially lead to a higher rate of arthrodesis, and preservation of a functional range of motion. However, comprehensive prospective studies detailing the outcomes, union rates, and complication profile of this specific procedure are still relatively scarce in the literature. ResearchGate - Lunate-capitate arthrodesis (2024)]. This study is designed to prospectively evaluate the efficacy and safety of lunocapitate fusion as a primary surgical treatment for SNAC wrist. The rationale is to provide robust clinical data that can solidify the role of LC fusion in the management algorithm of this condition.

Lunocapitate (LC) fusion has emerged as a promising salvage technique. By reducing the number of fusion sites compared to other procedures, it aims to achieve a higher union rate, reduce operative time, and better preserve wrist motion. However,comprehensive prospective data on its outcomes are still needed. This study will prospectively evaluate the efficacy and safety of lunocapitate fusion as a primary surgical treatment for SNAC wrist.

ELIGIBILITY:
Inclusion Criteria:

* 1- Age 18-60 years 2- symptomatic SNAC wrist failed conservative management.

Exclusion Criteria:

* 1- total wrist Arthritis 2-systemic arthropathy 3-Infected wrist

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-03-10 (Estimated)

PRIMARY OUTCOMES:
DASH SCORE | 12 month
Functional outcome measured by the DASH score at 12 months post-operation | 12 month

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27839956/